CLINICAL TRIAL: NCT07034313
Title: Rouen Study on Anxiety During Allergy Tests
Brief Title: Rouen Study on Anxiety
Acronym: ERATA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0241/OB; N° IDRCB : 2024-A02144-43 (Other: ANSM)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-01

CONDITIONS: Anxiety Disorder
Keywords: allergy test
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient benefiting from allergy tests

SUMMARY:
Allergy testing is necessary to confirm a diagnosis of allergy, whether food, respiratory, drug, or hymenoptera venom.

Although the vast majority of these tests are well tolerated, performing them carries a very low risk of inducing an allergic reaction in the patient, warranting continuous medical monitoring regardless of the allergy being investigated.

A severe reaction can be observed, largely during oral or intravenous reintroduction tests, in up to 15% of series for food allergies, and even less for drug allergies.

The perceived risk can vary between patients, and this subjective perception can be influenced by several factors, including personal experience, medical history, or access to information regarding allergy testing. Anxiety related to allergy testing can influence patient experience, but also test results.

DETAILED DESCRIPTION:
The assessment of this anxiety and understanding of the factors that influence it remain understudied, particularly in patients undergoing allergy testing. This study seeks to measure this anxiety and the factors that may influence it, in order to tailor personalized care for each patient.

This study will be conducted through the administration of a standardized questionnaire designed to measure the anxiety of patients undergoing allergy testing, as well as several parameters that may influence this anxiety, such as the prevalence of depression and anxiety disorders, and personality traits influenced by stress, using specific and validated scores.

This questionnaire will be administered to patients attending Rouen University Hospital for skin allergy testing and oral or intravenous provocation testing.

This descriptive study will focus on analyzing patients' perceptions and experiences without directly interfering with the medical procedures performed. Patients' perceptions and experiences will be collected using statements that will be rated on a Likert scale by the patients

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18 years old), of both sexes.
* Patient undergoing allergy testing (provocation or skin prick tests) at the Erik Satie Center during the inclusion period.
* Patient affiliated with a social security scheme
* Patient who has read and understood the information letter and does not object to participating in the study

Exclusion Criteria:

* Patient under guardianship or curatorship.
* Patient suffering from a psychological or sensory abnormality likely to prevent the patient from fully understanding the conditions required for participation in the study or to prevent the patient from giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing skin allergy testing
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Measure anxiety in patients undergoing allergy testing | 1 day
  The primary endpoint will be the visual analogue anxiety scale with a score ranging from 0 (total absence of anxiety) to 10 (maximum anxiety), before allergy testing is performed.

SECONDARY OUTCOMES:
Prevalence of anxiety disorders | 1 day
  Anxiety-depressive disorders will be assessed using the HAD (Hospital Anxiety and Depression scale) questionnaire, administered to patients included in the study.
Prevalence of anxiety disorders | 1 day
  Anxiety-depressive disorders will be assessed using the PSS (Perceived Stress Scale) questionnaire, administered to patients included in the study.
Patient care pathways | 1 day
  Information on the care pathway will be collected using closed (multiple choice) questions (general information).
Positivity rate of the various allergy tests | 1 day
  The results of the allergy tests will be studied by consulting the clinical file, and will be analyzed for their association with anxiety levels.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien SF FRANCHINA, Doctor, Principal Investigator — University Rouen Hospital
Locations (1):
- Service d'Allergologie, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.